CLINICAL TRIAL: NCT05372406
Title: Clinical Prediction Model and External Validation of Chronic Postsurgical Pain in Elders: Retrospective Analysis of A Multi-Center Prospective Database in China
Brief Title: Clinical Prediction Model and External Validation of Chronic Postsurgical Pain in Elders
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); First Affiliated Hospital of Guangxi Medical University (Other); Sun Yat-sen University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Peking University People's Hospital (Other); China-Japan Friendship Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Yanhong Liu, Deputy Chief of administration, Anesthesiology, Chinese PLA General Hospital
Other Study IDs: PLAGH-CPSP-001
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Chronic Postsurgical Pain
Keywords: elderly; Chronic Postsurgical Pain; Prediction; risk factors; Validation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group: elderly patients (aged ≥ 65 years) elderly patients undergo surgeries
  Interventions: Other: • no intervention
- external validation group: elderly patients (aged ≥ 65 years) elderly patients undergo surgeries
  Interventions: Other: • no intervention

INTERVENTIONS:
Other: • no intervention — • no intervention

SUMMARY:
This study will collect perioperative pain-related data of elderly patients in multi-centers. Analyzing these collected data to find the high-risk factors of chronic postsurgical pain in elderly patients and to establish an early-warning models of perioperative pain in elderly patients, so as to improve the ability of assessing the risks of postoperative pain in elderly patients and providing an early warning.

Based on the database, the investigators intend to explore:

* Perioperative risk assessment methods and early warning models for elderly patients;
* Practical, safe, and effective risk prevention and control system through subsequent studies.

DETAILED DESCRIPTION:
This study will collect perioperative pain-related data of elderly patients in multi-centers, including: preoperative general data, intraoperative anesthesia and surgical data, clinical laboratory data, postoperative pain and intervention, postoperative complications and quality of life. Analyzing these collected data to find the high-risk factors of chronic postsurgical pain in elderly patients and to establish an early-warning model of chronic postsurgical pain in elderly patients, so as to improve the ability of assessing the risks of chronic postsurgical pain in elderly patients and providing an early warning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic postsurgical pain (CPSP) CPSP was made based on the guidelines of the International Society for Pain (CPSP: ICD-11) as follows: Chronic postsurgical pain is chronic pain developing or increasing in intensity after a surgical procedure and persisting beyond the healing process, i.e. at least 3 months after surgery. The pain is either localised to the surgical field, projected to the innervation territory of a nerve situated in this area, or referred to a dermatome (after surgery/injury to deep somatic or visceral tissues). Other causes of pain including infection, malignancy etc. need to be excluded as well as pain continuing from a pre-existing pain problem. Dependent on type of surgery, chronic postsurgical pain often may be neuropathic pain.
* Geriatric surgical patients ≥65 years old

Exclusion Criteria:

* Patients in the central nervous system group were excluded from cardiac and neurosurgery, patients in the heart injury group were excluded from cardiac surgery, and patients who did not agree to participate in the study were excluded in all groups.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 7770 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pain trajectories after surgery (Numerical Rating Scale) | Up to 3 months postoperation
  Pain intensity was assessed using a numerical rating scale (NRS) from 0 to 10, with zero representing no pain and 10 representing worst imaginable pain. The worst pain intensity was then categorized into two groups: no or mild pain (NRS from 0 to 3) and moderate to severe pain (NRS from 4 to 10).
The Brief Pain Inventory-short form | Up to 3 months postoperation
  It measured pain location in the body; pain intensity on an 11-point numerical rating scale (NRS; 0 represents "no pain" and 10 the "worst pain imaginable"); analgesic intake; perception of analgesic relief; and pain interference with daily life on an 11-point NRS (0 "does not interfere and 10"completely interferes") indistinct dimensions (general activity, mood, walking, work, relations with others, sleep, and enjoyment of life). Higher scores represent higher levels of pain interference.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | within 30 days prior to surgery
  The PCS consists of 13 items, and each item is answered with a numeric value between 0 and 4; 0 corresponding to "not at all", and four corresponded to "all the time". Higher scores indicate a higher level of pain catastrophizing, the Chinese version of the PCS has demonstrated a good reliability and validity (Cronbach's alpha was 0.87 and the ICC was 0.97)
The trajectories of health related quality of life(HRQoL) | within 30 days prior to surgery , 1, 3, 7, 30, 90 days postoperation
  The trajectory of HRQoL is the vector of Utility values measured with EuroQol five-dimensional questionnaire(EQ-5D-5L)taken over 3 months(days 1, 3, 7, 30, 90；Day 0 is the day of surgery). The EQ-5D-5L measures health on five domains (mobility, self-care, usual activities, pain discomfort, and anxiety-depression), and the scores will be combined using Chinese general population weights to generate a single utility or index score. Utility values for the EQ-5D range from 1.00 to -0.391, where a score of 0 and 1 are regarded as equivalent to death and 'perfect health', respectively, and a score < 0 is considered as health state that is 'worse than death'.
The Hospital Anxiety and Depression Scale | within 30 days prior to surgery , Up to 3 months postoperation
  Comprised by 2 subscales used to measure anxiety and depression through 7 items each. Subscale scores range from 0 to 21 and result from the sum of each item (Likert scale ranging from 0 to 3). Higher scores correspond to higher levels of anxiety and depression.
FRAIL Scale | within 30 days prior to surgery ,Up to 3 months postoperation
  Frailty was assessed within 30 days prior to surgery using the FRAIL Scale assessment. The FRAIL Scale assessment is a validated 5-item scale comprising components from the Cardiovascular Health Frailty Index and Rockwood Scale.The five components measured include fatigue, resistance, ambulation, illness and loss of weight. The scale was dichotomized into two frailty categories based on prior literature on pain and frailty.16 Patients were classified as frail if they scored 3 or more on the 5-point scale and not frail if they scored below 3 .
Complications within 30 days after surgery | Up to 3 months postoperation
  Complications within 30 days after surgery will be classified using Clavien-Dindo Classification of Surgical Complications, ranging from Grade I(Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions) to Grade V(death of a patient).
Postoperative duration of stay in hospital | Up to 3 months postoperation
  The duration when patients stay in hospital after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Weidong, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided